CLINICAL TRIAL: NCT07231588
Title: Feasibility of an Oral 5 Strain Probiotic (PGC) for GI Toxicity Mitigation During Pelvic Radiation
Brief Title: Oral 5 Strain Probiotic for GI Toxicity Mitigation During Pelvic Radiation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Pendulum Therapeutics (Industry)
Responsible Party: Principal Investigator, Bailey Nelson, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCC-RT-25-02
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Radiation Injuries
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RT + Probiotic (Experimental): Pendulum Glucose Control (PGC) probiotic + Radiation Therapy Treatment
  Interventions: Biological: Pendulum Glucose Control (PGC)

INTERVENTIONS:
Biological: Pendulum Glucose Control (PGC) — Pendulum Glucose Control (PGC) WBF-038 - 2 capsules Orally with food. Once daily for 10 weeks

SUMMARY:
This research is to determine if an oral probiotic, Pendulum Glucose Control (PGC), can be safely given to patients during pelvic radiation therapy (RT). The researchers will study if the probiotics lessen gastrointestinal toxicity during pelvic radiation.

DETAILED DESCRIPTION:
The exact mechanism of GI symptoms is elusive, but there is sufficient data to suggest that the intestinal microbiome plays a role in radiation-induced GI injury. The investigators propose a pilot feasibility trial evaluating whether an oral 5 strain probiotic (PGC) can be safely and effectively administered during pelvic RT. PGC will be supplied by Pendulum Therapeutics. Pendulum has completed trials using PGC in non-cancer conditions [26]. The investigators hypothesize that oral supplementation with PGC for GI toxicity mitigation during pelvic radiation is feasible. The intervention will be considered feasible if probiotic tolerability and patient adherence are appropriate. An overall probiotic adherence rate of ≥ 80% by ≥ 70% of patients will be considered acceptable. If feasible, these results will support evaluation of toxicity mitigation in randomized subsequent Phase II/III trials of PGC supplementation during pelvic radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed malignancy for which the standard of care treatment is at least 30 Gy of pelvic RT to the pelvic lymph nodes.

   a. Eligible diagnoses include: i. Lower GI cancers (anal, rectal) ii. Gynecologic cancers (cervical, vulvar, vaginal, endometrial) iii. Prostate cancer with lymph node involvement
2. Age ≥18 years.
3. ECOG performance status ≤2 (or Karnofsky ≥60%, see Appendix A).
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with inflammatory bowel disease (IBD - such as Crohn's or Ulcerative Colitis).
2. Patients who are currently receiving any other investigational agents. Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI.
3. Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous, in the opinion of the Investigator.
4. Patients with a prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of the investigational regimen in the opinion of the Investigator.
5. Patients who have received previous radiation therapy to the pelvis at any time.
6. Patients who have not recovered from GI adverse events due to previous cancer therapy.
7. Patients with colostomy or ileostomy.
8. Pregnant women are excluded from this study because they cannot receive radiotherapy.
9. Known inulin intolerance or allergies or hypersensitivity to any of the components of PGC, including:

   1. Known hypersensitivity to >4 first-line antimicrobial therapies against Akkermansia muciniphila, Clostridium beijerinckii, Clostridium butyricum, Anaerobutyricum hallii: Penicillin, Piperacillin, Tetracycline, Amoxicillin, Ampicillin
   2. Known hypersensitivity to >4 first-line antimicrobial therapies against Bifidobacterium infantis Bi-26TM: Gentamicin, Kanamycin, Streptomycin, Tetracycline, Erythromycin, Clindamycin, Ampicillin, Vancomycin
10. Patients unable to swallow capsules.
11. Absolute Neutrophil Count (ANC) < 1500/uL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Pendulum Glucose Control (PGC) Probiotic Adherence Rate (PAR)- measured by pill counts | Week 6 and week 10
  1. To evaluate Pendulum Glucose Control (PGC) Probiotic Adherence Rate (PAR).
  a. To assess Probiotic Adherence Rate (PAR), pill counts will be conducted at week 6 and week 10.

SECONDARY OUTCOMES:
Physician-reported GI toxicity with the addition of PGC - measured by CTCAE v6 | Baseline, week 4, week 6 and week 10. Week 14 (safety visit)
  To assess physician-reported GI toxicity, AEs using CTCAE v6 will be collected at baseline, week 4, week 6 and week 10. This will also be assessed at the 30 day safety visit after patients discontinue the supplement.
Patient-reported GI toxicity with the addition of PGC measured by PRO-CTCAE | Baseline, week 4, week 6 and week 10. Week 14 (safety visit)
  To assess patient-reported GI toxicity, an EPIC Bowel and a customized PRO-CTCAE will be collected at baseline, week 4, week 6 and week 10. This will also be assessed at the 30 day safety visit after patients discontinue the supplement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided